CLINICAL TRIAL: NCT01295060
Title: PHASE IIIB, OPEN-LABEL, MULTICENTER STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF AN 84-MG OCTREOTIDE SUBCUTANEOUS HYDROGEL IMPLANT IN SUBJECTS WITH ACROMEGALY
Brief Title: Long-term Safety and Efficacy Study of Octreotide Implant in Patients With Acromegaly
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program was terminated for business reasons
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3332-301
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Acromegaly
Keywords: Acromegaly; Octreotide; IGF-1; Growth Hormone; Implant; Hydrogel
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Octreotide Implant (Experimental)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide — 84 mg Octreotide Implant

SUMMARY:
This is a long term study to evaluate the safety, tolerability and efficacy of an Octreotide Implant in patients that were previously treated with an Octreotide implant.

DETAILED DESCRIPTION:
Evaluation on the long-term safety and tolerability, including local tolerability of the implant site, of the 84-mg octreotide hydrogel implant in subjects with acromegaly who had been successfully treated with the 84-mg octreotide hydrogel implant in the Phase III study IP107-001.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the Extension Phase of Study IP107-001 and received at least one 84-mg octreotide hydrogel implant prior to enrollment OR previously enrolled in the Extension Phase of Study IP107-001 and currently taking lanreotide or octreotide.
* Subjects who have been successfully treated with the 84-mg octreotide hydrogel implant in Study IP107 001.
* In the opinion of the Investigator; subject has no unstable chronic medical conditions and no clinically significant findings that would preclude subject's participation in the study.
* Subjects must be able to communicate, provide and sign written informed consent, and be willing to participate and comply with study requirements.

Exclusion Criteria:

* Pituitary surgery less than 3 months prior to enrollment into this study
* Liver disease (eg, cirrhosis, chronic active or persistent hepatitis or persistent abnormalities of ALT, AST [level >2× normal] or direct bilirubin [level >1.5× normal])
* Unstable angina, sustained ventricular arrhythmias or heart failure (NYHA III and IV)
* Acute myocardial infarction within 3 months of Screening
* Uncontrolled diabetes defined as having an HbA1c ≥9%
* Symptomatic cholelithiasis
* History of drug or alcohol abuse
* Received any investigational drug or participated in another clinical trial except for study IP107 001 within 30 days of enrollment into this study
* Received radiotherapy for pituitary tumor or any radiotherapy above the neck at any time prior to enrollment into this study
* Receiving pegvisomant, dopamine agonist or other therapy in combination with somatostatin to control GH or IGF-1 levels prior to enrollment into this study
* History or presence of significant cardiovascular, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease, any other severe coexisting or, terminal systemic disease that limits life expectancy, or may interfere with the conduct of the study, or subjects who are incarcerated in penal institutions or are committed to mental institutions
* Women who are pregnant or lactating. For females of childbearing potential, a positive pregnancy test prior to enrollment, or an unwillingness to use accepted forms of reliable birth control for study duration (including bilateral tubal ligation, use of oral contraceptives, double barrier methods [diaphragm with spermicidal gel or condoms with contraceptive foam], Depo-Provera®, hormonal implants, partner vasectomy, and total abstinence). Pregnancy tests are not required (indicate "n/a") for males, or for females not of childbearing potential (post-menopausal with last menstrual period >1 year ago or total hysterectomy with bilateral oophorectomy)
* An unwillingness on the part of a male subject to abstain from sexual intercourse with pregnant or lactating women or an unwillingness to use a condom and spermicide and another form of contraception (eg, IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant until discharge from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Long term safety and tolerability of the Octreotide Implant | every 3 months for up to 2 years
  Subjects will be assessed every 3 months via adverse event reporting and examination of the implantation site

SECONDARY OUTCOMES:
Evaluate the long term efficacy of the Octreotide Implant | every 3 months for up to 2 years
  Patients will have GH and IGF-1 analyzed every 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Denver, Colorado
  - Chicago, Illinois
  - Baltimore, Maryland
  - Cleveland, Ohio
  - Portland, Oregon
  - Seattle, Washington